CLINICAL TRIAL: NCT00004884
Title: Randomized Phase II Study of Docetaxel/Gemcitabine vs. Docetaxel/Cisplatin in Metastatic or Locoregionally Advanced Pancreatic Carcinoma
Brief Title: Docetaxel and Gemcitabine Compared With Docetaxel and Cisplatin in Treating Patients With Metastatic or Locally Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: EORTC-40984; EORTC-40984
Record Dates: First submitted 2000-03-07; First posted 2004-05-03 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Pancreatic Cancer
Keywords: stage III pancreatic cancer; recurrent pancreatic cancer; adenocarcinoma of the pancreas; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Cisplatin; Docetaxel; Gemcitabine

INTERVENTIONS:
Drug: cisplatin
Drug: docetaxel
Drug: gemcitabine hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. It is not yet known whether docetaxel plus gemcitabine is more effective than docetaxel plus cisplatin in treating advanced pancreatic cancer.

PURPOSE: Randomized phase II trial to compare the effectiveness of docetaxel and gemcitabine with that of docetaxel and cisplatin in treating patients who have metastatic or locally advanced pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the efficacy of docetaxel and gemcitabine vs docetaxel and cisplatin in patients with metastatic or locoregionally advanced pancreatic cancer. II. Assess the toxicity, response rate, duration of response, time to progression, survival, performance status, and weight associated with these treatment regimens in these patients.

OUTLINE: This is a randomized, open label, multicenter study. Patents are randomized to one of two treatment arms. Arm I: Patients receive gemcitabine IV over 30 minutes on days 1 and 8 and docetaxel IV over 1 hour on day 8. Arm II: Patients receive docetaxel IV over 1 hour followed by cisplatin IV over 1 hour on day 1. Treatment is repeated every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients are followed every 6 weeks until disease progression, and then every 8 weeks until death.

PROJECTED ACCRUAL: Up to 82 patients (41 per arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed metastatic or locoregionally advanced (with metastatic lymph nodes) unresectable adenocarcinoma of the exocrine pancreas Bidimensionally measurable disease outside previously irradiated fields No CNS involvement or leptomeningeal disease

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: WHO 0-1 Life expectancy: Not specified Hematopoietic: WBC at least 3,000/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin less than 1.5 times the upper limit of normal (ULN) Renal: Creatinine no greater than ULN Other: No prior second malignancy in the past 10 years except carcinoma in situ of the cervix or basal or squamous cell carcinoma of the skin No psychological, familial, sociological, or geographical condition that precludes study compliance Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior immunotherapy Chemotherapy: No prior chemotherapy Endocrine therapy: Not specified Radiotherapy: Concurrent radiotherapy allowed if indicator lesions not included in irradiated field See Disease Characteristics Surgery: Not specified Other: No concurrent investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 1999-07; Primary Completion 2001-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Lutz, MD, Study Chair — Comprehensive Cancer Center Ulm at Universitaetsklinikum Ulm
Locations (19):
- Belgium (3):
  - Institut Jules Bordet, Brussels
  - Hopital Universitaire Erasme, Brussels
  - U.Z. Gasthuisberg, Leuven
- National Cancer Institute of Egypt, Cairo, Egypt
- France (3):
  - CHU Ambroise Pare, Boulogne-Billancourt
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif
- Germany (8):
  - Klinikum St. Marien, Amberg
  - Universitaetsklinik und Strahlenklinik - Essen, Essen
  - Klinikum der J.W. Goethe Universitaet, Frankfurt
  - Marien Hospital, Hagen
  - Hermann-Holthusen Institute for Radiotherapy, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Praxis Innere Medizin, Neustadt
  - Klinikum der Universitaet Ulm, Ulm
- Saint Laurentius Ziekenhuis, Roermond, Netherlands
- Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology, Warsaw, Poland
- Dokuz Eylul University School of Medicine, Izmir, Turkey (Türkiye)
- Beatson Oncology Centre, Glasgow, Scotland, United Kingdom

REFERENCES:
- [Result] Lutz MP, Van Cutsem E, Wagener T, Van Laethem JL, Vanhoefer U, Wils JA, Gamelin E, Koehne CH, Arnaud JP, Mitry E, Husseini F, Reichardt P, El-Serafi M, Etienne PL, Lingenfelser T, Praet M, Genicot B, Debois M, Nordlinger B, Ducreux MP; European Organisation for Research and Treatment of Cancer Gastrointestinal Group. Docetaxel plus gemcitabine or docetaxel plus cisplatin in advanced pancreatic carcinoma: randomized phase II study 40984 of the European Organisation for Research and Treatment of Cancer Gastrointestinal Group. J Clin Oncol. 2005 Dec 20;23(36):9250-6. doi: 10.1200/JCO.2005.02.1980. PMID 16361622
- [Result] Lutz MP, Ducreux M, Wagener T, et al.: Docetaxel/gemcitabine or docetaxel/cisplatin in advanced pancreatic carcinoma: a randomized phase II study of the EORTC-GI group. [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-498, 2002.